CLINICAL TRIAL: NCT06187051
Title: FEVAR or Open Repair to Treat Type 1 Endoleak : A French Multicentric Study
Brief Title: Type 1 Endoleak : Fenestrated Custom Made Endograft (FEVAR) Versus Open Surgery Explantation (OSR) : What's the Best
Status: Completed | Type: Observational
Sponsor: University Paul Sabatier of Toulouse (Other)
Responsible Party: Principal Investigator, Aurélien Hostalrich, Clinical Professor, University Paul Sabatier of Toulouse
Other Study IDs: Type 1 endoleak : FEVAR vs OSR
Record Dates: First submitted 2023-12-15; First posted 2024-01-02 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2024-01

CONDITIONS: Aorta Aneurysm
MeSH Terms: conditions — Aortic Aneurysm | interventions — Endovascular Aneurysm Repair; Device Removal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patient presenting a type 1A endoleak after EVAR treated by relining with FEVAR
  Interventions: Device: FEVAR
- Patient presenting a type 1A endoleak after EVAR treated by explantation of the EVAR
  Interventions: Device: Explantation

INTERVENTIONS:
Device: FEVAR — Relining the EVAR with FEVAR
  Groups: Patient presenting a type 1A endoleak after EVAR treated by relining with FEVAR
Device: Explantation — open surgery to explant the previous EVAR
  Groups: Patient presenting a type 1A endoleak after EVAR treated by explantation of the EVAR

SUMMARY:
Proximal type 1A endoleak is a worrying complication after endovascular repair of an abdominal aortic aneurysm (EVAR). The ideal solution is not obvious between relining by FEVAR and endograft explantation.

A retrospective french multicentric study was performed between 2010 and 2023 to compare the outcomes and the efficiency of both technics and propose a decision algorithm for the management of type 1A endoleak after EVAR.

ELIGIBILITY:
Inclusion Criteria:

* Type 1A endoleak after EVAR

Exclusion Criteria:

* no

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient presenting a type 1A endoleak after EVAR for AAA during the follow up
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2010-01-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Post operative mortality | day 30 post operative
  Patient death after the treatment of type 1A endoleak
Major adverse cardiovascular event (MACE) post operative | day 30 post operative
  Patient presenting after surgery a composite score (MACE) including
  * nonfatal stroke,
  * nonfatal myocardial infarction
  * cardiovascular death
Redo surgery after type 1A endoleak surgery | 30 day, 6 months, 12 months, 24 months
  Reintervention after FEVAR or explantation surgery

SECONDARY OUTCOMES:
Efficiency of the treatment | 30 day, 6 months, 12 months, 24 months
  No reintervention after open surgery or Thrombosis of the aneurysmal sac after FEVAR